CLINICAL TRIAL: NCT07388017
Title: High Resolution Thermographic Imaging as a Diagnostic Aid in Paediatric Infections of Bones, Joints, and Soft Tissues
Brief Title: Infrared Thermography for Diagnosis of Musculoskeletal Infections
Status: Recruiting | Type: Observational
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SCH-2913
Record Dates: First submitted 2025-02-18; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-03

CONDITIONS: Musculoskeletal Infection; Septic Arthritis; Osteomyelitis/Septic Arthritis
MeSH Terms: conditions — Arthritis, Infectious; Osteomyelitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic Arthritis: Patients are stratified into two arms. If the participant is admitted with septic arthritis they will be prepared to be taken to theatres to have routine surgery. After the patients is in the theatre under general anaesthesia and immediately prior to surgery the research team will perform the study intervention. This is using a High Resolution Thermal Imaging camera to take an image of the infected area.
  Interventions: Device: High Resolution Thermal Imaging
- Non-Emergent Musculoskeletal Infection: Patients are stratified into two arms. If the participant is admitted with a non emergent MSK infection, the patient will be prepared to have an MRI scan. Immediately prior to the MRI scan, the research team will perform the study intervention. This is using a High Resolution Thermal Imaging camera to take an image of the infected area.
  Interventions: Device: High Resolution Thermal Imaging

INTERVENTIONS:
Device: High Resolution Thermal Imaging — A HRTI camera is a non-invasive medical device that will be utilised on patients that present in ED with an MSK infection. The goal of this intervention is to answer the following:
  Can combined HRTI and blood tests provide a higher diagnostic reliability than HRTI on its own? Can combined HRTI and artificial intelligence (AI) provide a timelier (as compared to existing modalities) detection of bone, joint and soft tissue infection thus allowing a more effective treatment? What are patients views and feedback for the new HRTI method?

SUMMARY:
This is a pilot proof of feasibility study to explore the efficacy of High Resolution Infrared Thermographic Imaging (HRTI) to assist with the detection of musculoskeletal infections in children. In HRTI, a sensitive thermal camera is used to capture the temperature profile of the suspected infected body region in the form of images. In this study, a 10-second video will be recorded to allow dynamic monitoring. The resulting video will be processed and interpreted to determine whether there is a musculoskeletal infection.

Bone, joint and soft tissue infections can be caused by bacteria which can enter the body through accidental injuries, or because of surgery or implants. Once in the body, they circulate through the bloodstream until they reach a bone, joint, or muscle, multiply and cause infection. These conditions can cause significant complications in children and adults and can even result in death if untreated.

Infections of the bone, called osteomyelitis can inhibit bone growth in children. As a result, children who have suffered from osteomyelitis may require extensive treatment later in childhood. While osteomyelitis accounts for only 1% of childhood hospital admissions, its incidence in children has increased in recent decades. This is associated with an increase in the prevalence of antibiotic resistant bacteria such as MRSA.

Infections of the joint, called septic arthritis, is an emergency condition that requires prompt diagnosis and treatment. Long delays in diagnosis and surgical drainage of the joint may lead to irreversible damage to the cartilage and bone destruction.

There is currently a need for improved technologies to screen for and monitor bone, joint, and soft tissue infections. Plain radiographs appear normal in the first 7 to 10 days of osteomyelitis. Magnetic resonance imaging (MRI) is the most sensitive modality for diagnosing osteomyelitis. However, MRI scans are costly their accessibility is limited, plus the scan can take 30 minutes to perform. As the child needs to be still during the scan, sedation is required.

Infrared thermal imaging is a harmless, cost effective and rapid scanning method that has proven industrial applications such as condition monitoring of machineries and fault findings. There has also been extensive interest in utilising and this technology for medical diagnosis and monitoring. This study builds on our earlier work that used HRTI to detect inflammation in the abdomen in infants. This technology may allow timelier and more cost-effective diagnosis of the condition. Sheffield Children's Hospital and Sheffield Hallam University collaborate in conducting the study.

The study will involve recruiting 30 patients at Sheffield Children's Hospital with suspected infection of either bone, joint or soft tissue. They will have their HRTI recorded and processed to follow up the study's research questions. The findings from the study will not alter the routine medical treatments of the patients and participation is voluntary.

ELIGIBILITY:
Inclusion Criteria:

* Children and young people from neonates to 15 years of age:
* With clinical suspicion of a primary MSK infection (irrespective of location or aetiology), as defined by presenting symptoms, physical examination and bloodwork performed by a qualified clinician.
* Presenting to Sheffield Children's Hospital via A&E or referral from another hospital.
* Who are able to interpret the information given in the information sheet/assent form on paper in English (with the exception of children under the age of 3 years who are not required to assent.)
* With at least 1 competent legal guardian who is capable of legally consenting, and interpreting the information given in the information sheet in English.
* Where a medical doctor involved in their care has agreed that their participation in the study will not negatively impact on their treatment outcome

Exclusion Criteria:

* - Have a secondary MSK infection.
* Are severely ill or need urgent/critical attention or have comorbid conditions that will complicate their care, as decided by a medical doctor involved in their treatment.
* Patients with conditions including but not limited to leukaemia, hyper/hypothyroidism, diabetes mellitus or any other condition that affects their basal metabolic rate/body temperature.
* Amputees where the amputated region is contralateral to the region of suspected infection.
* Have received an a priori diagnosis or have already undergone any investigation. This includes patients admitted for a recurrence/exacerbation of recently diagnosed MSK infection.
* Any patient where the medical team responsible for their treatment raises concerns that HRTI could negatively impact their treatment outcome.
* The patient, or their legal guardian(s) do not consent or assent/withdraw consent or assent/ or are not able to consent or assent for any reason. (Eg. The patient/guardian(s) are non-English speakers or have disabilities impairing their understanding of the study.)

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paediatric patients ages 0-15 presenting to Sheffield Children's Hospital with a suspected primary muscoloskeltal infection
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Thermal profile variability in affected and contralateral region of interest. | Admission to hospital (Day 1)
  On admission (Day 1), thermal images of the affected and contralateral limbs are obtained. This generates a thermal profile through which the temperature (°C) can be extracted. A region of interest is drawn around the suspected anatomical zone of the infection. This outcome measure will compare differences in the temperature (°C) of the affected and contralateral region of interest. This will include the mean temperature difference and the hottest and coldest spots in each zone, respectively.

SECONDARY OUTCOMES:
Erythrocyte Sedimentation rate (ESR) | On admission (day 1)
  On admission (DAY 1) blood will be drawn and ESR will be recorded in millimeters per hour (mm/hr)
C-reactive protein (CRP) | On admission (Day 1)
  On admission (DAY 1), blood will be drawn and CRP will be measured in milligrams per litre (mg/L).
White blood cell count (WBC) | On admission (day 1)
  On admission (DAY 1), bloods will be drawn and the white blood cell count (x10^9/L) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Children's NHS Foundatin Trust, Sheffield, South Yorkshire, United Kingdom